CLINICAL TRIAL: NCT01524900
Title: Observational Study Assessing the Safety, Efficacy and Treatment Adherence of Nevirapine Extended Release (Combined With Other Antiretroviral Drugs) in HIV Infected Patients in Daily Clinical Practice
Brief Title: Observational Study of Nevirapine Extended Release in Human Immunodeficiency Virus (HIV) Patients in Daily Clinical Practice
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1550
Record Dates: First submitted 2012-01-17; First posted 2012-02-02 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- nevirapine extended release

SUMMARY:
This Post Marketing Surveillance study will be performed as an open-label, prospective, non-interventional, uncontrolled study in Human immunodeficit Virus-1 (HIV-1) infected patients. Data will only be documented in patients for whom a pharmacotherapy with nevirapine extended release is initiated. Both anti-retroviral therapy (ART) naïve patients and pre-treated patients switching from nevirapine immediate release or other anti-retroviral therapy (ART) will be included in the study. The decision to initiate treatment with nevirapine extended release is independent of this study and is based entirely on individual patient need and the judgement of the treating physician. The aim of the study is to assess the safety and efficacy and treatment adherence of nevirapine extended release in HIV-1 infected patients in routine clinical practice. It is planned to document five visits for each patient over a twenty four week observational period.

DETAILED DESCRIPTION:
Study Design:

non-interventional uncontrolled observational study

ELIGIBILITY:
Inclusion criteria:

1. HIV-1 infected male and female 18 years and above;
2. anti-retroviral therapy (ART) naive and pre-treated patients switching from a nevirapine immediate release or other ART.

Exclusion criteria:

Consistent with the current VIRAMUNE prolonged release SPC.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV-1 infected patients
Sampling Method: Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- Austria (6):
  - Boehringer Ingelheim Investigational Site 6, Graz
  - Boehringer Ingelheim Investigational Site 5, Salzburg
  - Boehringer Ingelheim Investigational Site 1, Vienna
  - Boehringer Ingelheim Investigational Site 2, Vienna
  - Boehringer Ingelheim Investigational Site 3, Vienna
  - Boehringer Ingelheim Investigational Site 4, Wels
- Poland (14):
  - Boehringer Ingelheim Investigational Site 7, Bialystok
  - Boehringer Ingelheim Investigational Site 8, Bialystok
  - Boehringer Ingelheim Investigational Site 10, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 9, Bydgoszcz
  - Boehringer Ingelheim Investigational Site 11, Chorzów
  - Boehringer Ingelheim Investigational Site 12, Chorzów
  - Boehringer Ingelheim Investigational Site 13, Gdañsk
  - Boehringer Ingelheim Investigational Site 14, Gdañsk
  - Boehringer Ingelheim Investigational Site 15, Gdañsk
  - Boehringer Ingelheim Investigational Site 16, Krakow
  - Boehringer Ingelheim Investigational Site 17, Krakow
  - Boehringer Ingelheim Investigational Site 18, Poznañ
  - Boehringer Ingelheim Investigational Site 19, Wroc£aw
  - Boehringer Ingelheim Investigational Site 20, Wroc£aw
- Romania (33):
  - Boehringer Ingelheim Investigational Site 50, Bacau
  - Boehringer Ingelheim Investigational Site 51, Brasov
  - Boehringer Ingelheim Investigational Site 52, Brasov
  - Boehringer Ingelheim Investigational Site 53, Brasov
  - Boehringer Ingelheim Investigational Site 21, Bucharest
  - Boehringer Ingelheim Investigational Site 22, Bucharest
  - Boehringer Ingelheim Investigational Site 23, Bucharest
  - Boehringer Ingelheim Investigational Site 24, Bucharest
  - Boehringer Ingelheim Investigational Site 25, Bucharest
  - Boehringer Ingelheim Investigational Site 26, Bucharest
  - Boehringer Ingelheim Investigational Site 27, Bucharest
  - Boehringer Ingelheim Investigational Site 28, Bucharest
  - Boehringer Ingelheim Investigational Site 29, Bucharest
  - Boehringer Ingelheim Investigational Site 30, Bucharest
  - Boehringer Ingelheim Investigational Site 31, Bucharest
  - Boehringer Ingelheim Investigational Site 32, Bucharest
  - Boehringer Ingelheim Investigational Site 33, Bucharest
  - Boehringer Ingelheim Investigational Site 34, Bucharest
  - Boehringer Ingelheim Investigational Site 35, Bucharest
  - Boehringer Ingelheim Investigational Site 36, Bucharest
  - Boehringer Ingelheim Investigational Site 37, Bucharest
  - Boehringer Ingelheim Investigational Site 38, Bucharest
  - Boehringer Ingelheim Investigational Site 39, Bucharest
  - Boehringer Ingelheim Investigational Site 40, Bucharest
  - Boehringer Ingelheim Investigational Site 41, Bucharest
  - Boehringer Ingelheim Investigational Site 42, Bucharest
  - Boehringer Ingelheim Investigational Site 43, Bucharest
  - Boehringer Ingelheim Investigational Site 44, Bucharest
  - Boehringer Ingelheim Investigational Site 46, Constanța
  - Boehringer Ingelheim Investigational Site 47, Constanța
  - Boehringer Ingelheim Investigational Site 48, Constanța
  - Boehringer Ingelheim Investigational Site 45, Giurgiu
  - Boehringer Ingelheim Investigational Site 49, Ploieşti

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 387 patients started treatment.
Groups:
- Treatment-naive Patients: Patients who were not pretreated with HIV therapy
- Patients Switching From Nevirapine IR: Patients switching from nevirapine immediate release (IR).
- Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL: Patients switching from a virologically effective treatment regimen (i.e. due to intolerance) other than nevirapine IR, with a baseline viral load ≤ 50 copies/mL.
- Pretreated Patients, Baseline Viral Load >50 Copies/mL: Patients switching from a virologically ineffective treatment regimen (i.e. due to intolerance) other than nevirapine IR, with a baseline viral load > 50 copies/mL.
- Patients With Baseline Viral Load Not Documented: Patients with no documented information about the baseline viral load.
Period: Overall Study
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Started | 49 | 246 | 30 | 22 | 40
Completed | 43 | 232 | 29 | 21 | 40
Not Completed | 6 | 14 | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 12 | 1 | 0 | 0
Not completed — Other reason than stated above | 1 | 1 | 0 | 0 | 0
Not completed — No reason documented | 2 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients from the Treated Set (TS): This patient set includes all HIV-1 infected patients who were dispensed Viramune® and were documented to have taken at least one dose of Viramune®and of a antiretroviral combination partner.
Groups:
- Pretreated Patients, Baseline Viral Load>50 Copies/mL: Patients switching from a virologically ineffective treatment regimen (i.e. due to intolerance) other than nevirapine IR, with a baseline viral load > 50 copies/mL.
- Total: Total of all reporting groups
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load>50 Copies/mL | Patients With Baseline Viral Load Not Documented | Total
Number analyzed (Participants) | 49 | 246 | 30 | 22 | 40 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (9.9) | 39.8 (13.8) | 38.1 (11.1) | 33.1 (10.4) | 37.4 (13.2) | 38.5 (13.1)
Gender [Number; unit: participants] — There are two patients with missing gender information, one in the group of the patients switching from nevirapine IR and one in the group of pretreated patients with HIV RNA>=50.
  participants
    Female | 8 | 90 | 11 | 7 | 19 | 135
    Male | 41 | 155 | 19 | 14 | 21 | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Non-serious Adverse Events, Serious Adverse Events, and Non-serious and Serious Adverse Events Leading to Treatment Discontinuation
Description: The primary endpoint is to evaluate the safety of a highly active antiretroviral therapy (HAART) that includes nevirapine extended release in routine clinical practice which is to assess the number of patients reporting non-serious adverse events (nSAEs), the number of patients with serious adverse events (SAE), the number of patients with non-serious adverse events leading to treatment discontinuation, and the number of patients with serious adverse events leading to discontinuation.
Time Frame: up to 72 weeks
Population: Patients from TS.
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 49 | 246 | 30 | 22 | 40
participants
  Patients reporting non-serious adverse events | 0 | 4 | 0 | 0 | 0
  Patients with serious adverse events | 0 | 2 | 0 | 0 | 0
  Patients with nSAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0
  Patients with SAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Patients With Virologic Response at Week 24 (Viral Load <50 Copies/mL)
Description: Virologic response is defined as confirmed Human Immunodeficiency Virus (HIV) viral load of < 50 copies/mL (at two consecutive measurements after baseline) up to week 24 and without subsequent rebound or change of anti-retroviral (ARV) therapy up to week 24. A rebound is defined as two consecutive measurements of viral load (VL) ≥ 50 copies/mL, at least two weeks apart, after two consecutive measurements of VL< 50 copies/mL. A change of ARV therapy is defined as a permanent discontinuation of nevirapine extended release, addition of new ARV drugs, or alteration in background therapy. A change in the background therapy due to toxicity or intolerance is not considered as treatment failure. If no follow-up viral load was available the virologic response is Missing.
Time Frame: 24 weeks
Population: Patients from the Full analysis set (FAS): This patient set includes all patients in the treated set who have analysable data in at least one efficacy endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 40 | 223 | 29 | 21 | 37
participants
  Virologic response | 21 | 150 | 15 | 3 | 11
  No virologic response | 3 | 10 | 1 | 2 | 1
  Missing | 16 | 63 | 13 | 16 | 25

3. Secondary Outcome: Change in CD4+ Cell Count From Baseline to Week 24
Description: The change in the Cluster of differentiation 4 (CD4+) cell count from baseline after 24 weeks was calculated by subtracting the baseline value from the value after 24 weeks. Therefore, a positive change represents an increase in CD4+ cell count.
Time Frame: baseline and week 24
Population: Patients from FAS with documented CD4+ at baseline and after 24 weeks.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 23 | 156 | 22 | 13 | 27
cells/mm^3 | 19.6 (347.8) | 98.9 (199.7) | 73.5 (152.2) | 31.2 (148.4) | 135.9 (583.5)

4. Secondary Outcome: Change in Morisky Medication Adherence Scale Score From Baseline to 24 Weeks
Description: The Morisky Medication Adherence scale (MMAS-8 scale) is a recognized indicator of medication adherence, consisting of 8 questions with a sum score ranging between 0 and 8 points. The higher score indicates higher adherence to the prescribed therapy recommendation. It has been agreed that the score of 8 could be categorized as having high adherence, score between 6 and 7 as medium adherence and scores of 5 and less as low adherence. The change is presented as the score after 24 weeks minus the score at baseline. Therefore, a positive change score reflects an improvement in the adherence.
Time Frame: baseline and week 24
Population: Patients from FAS with documented MMAS-8 score at baseline and after 24 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 17 | 205 | 28 | 21 | 33
units on a scale | 0.3 (1.1) | 0.4 (1.2) | 0.7 (1.2) | 0.8 (2.1) | -0.1 (1.2)

5. Secondary Outcome: Number of Patients Reporting Once Daily Nevirapine Intake More Convenient Than Twice Daily Formulation
Description: The number of patients reporting that they find the once daily nevirapine intake more / very much more convenient than the twice daily formulation.
Time Frame: 24 weeks
Population: Patients from FAS
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load >50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 40 | 223 | 29 | 21 | 37
participants
  Once daily intake is more convenient | 4 | 41 | 6 | 4 | 7
  Once daily intake is very much more convenient | 29 | 105 | 17 | 14 | 26

6. Primary Outcome: Number of Patients Reporting Rash of Any Severity
Description: Number of patients reporting rash of any severity as adverse event
Time Frame: up to 72 weeks
Population: Patients TS
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load>50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 49 | 246 | 30 | 22 | 40
participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Patients Reporting Hepatic Events
Description: Number of patients reporting hepatic events either as adverse event (AE) or as laboratory abnormality of Grade 1 to Grade 4 in aspartate aminotransferase (AST), alanine transaminase (ALT), Gamma-Glutamyl-Transferase (Gamma-GT) and bilirubin.
Time Frame: up to 72 weeks
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load>50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 49 | 246 | 30 | 22 | 40
participants
  Hepatic events reported as AE | 0 | 0 | 0 | 0 | 0
  Abnormality in AST | 1 | 3 | 1 | 4 | 1
  Abnormality in ALT | 11 | 22 | 7 | 9 | 8
  Abnormality in Gamma-GT | 11 | 64 | 7 | 5 | 4
  Abnormality in Bilirubin | 4 | 3 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Groups:
- Treatment-naïve Patients: Patients who were not pretreated with HIV therapy
- Pretreated Patients, Baseline Viral Load > 50 Copies/ML: Patients switching from a virologically ineffective treatment regimen (i.e. due to intolerance) other than nevirapine IR, with a baseline viral load > 50 copies/mL.
Arm/Group | Treatment-naïve Patients | Patients Switching From Nevirapine IR | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/ML | Pretreated Patients, Baseline Viral Load > 50 Copies/ML | Patients With Baseline Viral Load Not Documented
Serious Adverse Events (participants affected / at risk) | 0/49 | 2/246 | 0/30 | 0/22 | 0/40
Other Adverse Events (participants affected / at risk) | 0/49 | 0/246 | 0/30 | 0/22 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naïve Patients (N=49) | Patients Switching From Nevirapine IR (N=246) | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/ML (N=30) | Pretreated Patients, Baseline Viral Load > 50 Copies/ML (N=22) | Patients With Baseline Viral Load Not Documented (N=40)
Coronary artery disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.